CLINICAL TRIAL: NCT01983904
Title: Therapeutic Brain Stimulation for Refractory Depression
Brief Title: DBS for Treatment Resistant Depression
Acronym: CRIO-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Zelma Kiss, Associate Professor, Neurosurgery; Director Clinician Investigator Program, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-20948
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Major depressive disorder (MDD); Bi-polar disorder (BP)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long Pulse Width (Experimental): deep brain stimulation with short & long pulse width
  Interventions: Device: deep brain stimulation with short & long pulse width
- Short Pulse Width (Experimental): deep brain stimulation with short & long pulse width
  Interventions: Device: deep brain stimulation with short & long pulse width

INTERVENTIONS:
Device: deep brain stimulation with short & long pulse width — surgical implantation for bilateral electrodes and stimulation using short and long pulse width

SUMMARY:
The purpose of this study is to examine the effects of sub-callosal cingulate (SCC) deep brain stimulation (DBS) in patients with treatment resistant depression (TRD).

The working hypotheses are that long pulse-width DBS applied to the SCC region will lead to improvements in TRD patients, and specific neuroimaging biomarkers will correlate with response to DBS; the functional recovery will be enhanced with concurrent cognitive behavioural therapy (CBT).

DETAILED DESCRIPTION:
The aim is to collect data on prediction, optimization and augmentation of DBS for TRD and develop tools for DBS surgery. It is a biological pilot study designed to provide informative data for future work.

ELIGIBILITY:
Inclusion Criteria:

* age 20-70
* diagnosis of major depressive (MDD)or bipolar disorder(BP)determined independently by 2 study psychiatrists
* current major depressive episode of >1 year duration, treatment-resistant (meaning failure to respond to 4 different classes of antidepressants, including augmentation or combination strategies with lithium, atypical antipsychotics, anticonvulsants, antidepressants, evidence-based psychotherapy, CBT, or electroconvulsive treatment despite adequate dosage, duration and compliance)
* minimum score of 20 (out of 52) on the 17 item Hamilton Depression Rating Scale (HDRS)
* resident of Alberta, Canada, covered by Alberta Health

Exclusion Criteria:

* other Axis I psychiatric disorders including schizophrenia, psychosis, active suicidal ideation over previous 6 months
* cerebrovascular risk factors, previous stroke, head injury and neurodegenerative disorders, pregnancy, medical and general contraindications for DBS surgery (e.g. cardiac pacemaker/defibrillator)
* age >70
* diabetes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale | 6 and 12 months post-operatively
  change in HDRS from baseline before surgery: rates of remission (defined as an HDRS score <8 at 6 and 12 months) and response (defined as >50% reduction in HDRS)

SECONDARY OUTCOMES:
Change from baseline on Illness Density Index, Montgomery-Asberg Depression Rating Scale and Hamilton Anxiety Scale, Positive and Negative Affect Scale, Clinical Global Impression of Change, GAF< SAs, NAS, Q-LES-Q-SF & neuropsychological tests | 6 and 12 months post operatively
  change in MADRS score from baseline before surgery to 6 and 12 months post operatively
Post Cognitive Behavioural Therapy Scores | 15 months post operatively
  Changes in primary and secondary measures from pre-CBT scores will be used

CONTACTS AND LOCATIONS:
Overall Officials: Zelma H Kiss, MD PhDFRCSC, Principal Investigator — University of Calgary, Department of Clinical Neurosciences; Rajamannar Ramasubbu, MD MRCP FRCP, Principal Investigator — University of Calgary, Department of Psychiatry
Locations (1):
- University of Calgary & Alberta Health Services, Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Ramasubbu R, Brown EC, Mouches P, Moore JA, Clark DL, Molnar CP, Kiss ZHT, Forkert ND. Multimodal imaging measures in the prediction of clinical response to deep brain stimulation for refractory depression: A machine learning approach. World J Biol Psychiatry. 2024 Mar;25(3):175-187. doi: 10.1080/15622975.2023.2300795. Epub 2024 Jan 17. PMID 38185882
- [Derived] Ramasubbu R, Clark DL, Golding S, Dobson KS, Mackie A, Haffenden A, Kiss ZH. Long versus short pulse width subcallosal cingulate stimulation for treatment-resistant depression: a randomised, double-blind, crossover trial. Lancet Psychiatry. 2020 Jan;7(1):29-40. doi: 10.1016/S2215-0366(19)30415-8. PMID 31860455